CLINICAL TRIAL: NCT01746875
Title: Pigment Epithelium Detachment - a Prospective Clinical Study. PED-study.
Brief Title: A Study Testing if Medicine Can Make Pigment Epithelium Detachments Regress and Stabilize the Vision in Eyes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: treatment effects not as desired
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012/1743
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Macular Degeneration; Retinal Detachment
Keywords: Angiogenesis inhibitors; Photochemotherapy; Vascular Endothelium Growth Factors; Aflibercept
MeSH Terms: conditions — Macular Degeneration; Retinal Detachment | interventions — aflibercept; Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): aflibercept intravitreal injections, 2.0 mg monthly x 3 doses, then injections as needed based on recurrence of activity on OCT. If no effect of the treatment; aflibercept intravitreal injections, 2.0 mg x 3 doses is repeated, then injections as needed based on recurrence of activity on OCT. If no effect of the treatment; verteporfin photo dynamic therapy.
  Interventions: Drug: Aflibercept; Drug: Verteporfin
- Observation (No Intervention)

INTERVENTIONS:
Drug: Aflibercept — 2.0 mg monthly x 3 doses, then as needed based on recurrence of activity on OCT. If no effect after the initial 3 doses; 2.0 mg monthly x 3 doses is repeated.
  Arms: Treatment
Drug: Verteporfin — given if aflibercept does not have any effect. Verteporfin photodynamic therapy is given in combination with aflibercept and triamcinolone. The treatment can be repeated after 3 month.
  Arms: Treatment

SUMMARY:
The purpose of this study is to determine treatment effects in patients with retinal pigment epithelium detachment (PED) in relation to Age Related Maculopathy (AMD). Patients with newly diagnosed PED without choroidal neovascularisations (CNV), will be randomized to either treatment or observation. The treatment group will first be given injections with anti Vascular Endothelium Growth Factor (anti-VEGF). If the injections do not have any effect, Verteporfin Photodynamic Therapy (PDT) will be given. All patients will be followed for a period of 2 years. It is hypothesized that treatment stops the progression of the disease and stabilizes the vision in this subgroup of patients with AMD.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 50 years
* Pigment epithelium detachment in an eye not earlier treated with anti-VEGF or verteporfin PDT.
* ETDRS Best Corrected Visual acuity 20/32 - 20/400

Exclusion Criteria:

* Prior treatment with verteporfin, or external-beam radiation therapy, or transpupillary thermotherapy, Previous subfoveal focal laser photocoagulation involving the foveal center, History of vitrectomy, submacular surgery, or other surgical intervention for AMD.
* CNV, Subfoveal fibrosis or atrophy in study eye.
* Concurrent eye disease in the study eye that could compromise visual acuity (e.g., diabetic retinopathy, advanced glaucoma) or require medical or surgical intervention during the study. Active intraocular inflammation in the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Mean change in visual acuity from baseline to 24 months | 24 months
  Best corrected visual acuity (BCVA) on the Early Treatment for Diabetic Retinopathy Study (ETDRS) chart at 4 meters will be compared

SECONDARY OUTCOMES:
Visual acuity from baseline to 6 months | 6 months
  BCVA on ETDRS will be compared from baseline to 6 months
Visual acuity from baseline to 12 months | 12 months
  BCVA on ETDRS will be compared from baseline to 12 months
Safety | 24 months
  Incidence and severity of ocular and non-ocular adverse events will be evaluated through 24 months
Change in Optical Coherence Tomography (OCT) measurements from baseline through 24 months | 24 months
  Change in OCT Central Retinal Thickness (CRT) and Volume of PED from baseline through 24 months
Development of choroidal neovascularisations (CNV) | 24 months
  Development of CNV seen with OCT, fluorescein and indocyanine green imaging

CONTACTS AND LOCATIONS:
Overall Officials: Tor Elsaas, Prof. MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of Neuroscience, NTNU, Trondheim, Norway